CLINICAL TRIAL: NCT06667687
Title: A Phase 1 First-In-Human Study Evaluating Safety, Pharmacokinetics, and Efficacy of ABBV 291 as Monotherapy and in Combination in Non-Hodgkin's Lymphoma
Brief Title: Study to Evaluate Adverse Events, Change in Disease Activity, and How Intravenously Infused ABBV-291 Moves Through the Body in Adult Participants With Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-893; 2024-512586-13-00 (Other: EU CT)
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphomas; Diffuse Large B-Cell Lymphoma; Mantle Cell Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Waldenstroms Macrogloulinemia; Germinal Center B-cell; Activated B-Cell; NHL; DLBCL; MCL; FL; MZL; WM; GCB; ABC; Cancer; ABBV-291
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Escalation: Non-Hodgkin Lymphoma (NHL) ABBV-291 (Experimental): Participants with relapsed/refractory (R/R) B-cell non-Hodgkin lymphoma (NHL), except chronic lymphocytic leukemia (CLL), will receive escalating doses of ABBV-291, as part of the 74 month study duration.
  Interventions: Drug: ABBV-291
- Expansion: Diffuse Large B-Cell Lymphoma (DLBCL) ABBV-291 (Experimental): Participants with R/R DLBCL will receive the recommended Phase 1 expansion dose (RP1ED) of ABBV-291, as part of the 74 month study duration.
  Interventions: Drug: ABBV-291
- Expansion: Follicular Lymphoma (FL) ABBV-291 (Experimental): Participants with R/R FL will receive the RP1ED of ABBV-291, as part of the 74 month study duration.
  Interventions: Drug: ABBV-291
- Optimization: Mantle Cell Lymphoma (MCL) ABBV-291 Dose A (Experimental): Participants with R/R MCL will receive the dose A of ABBV-291, as part of the 74 month study duration.
  Interventions: Drug: ABBV-291
- Optimization: MCL ABBV-291 Dose B (Experimental): Participants with R/R MCL will receive the dose B of ABBV-291, as part of the 74 month study duration.
  Interventions: Drug: ABBV-291
- Optimization: MCL ABBV-291 Dose C (Experimental): Participants with R/R MCL will receive the dose C of ABBV-291, as part of the 74 month study duration.
  Interventions: Drug: ABBV-291

INTERVENTIONS:
Drug: ABBV-291 — Intravenous Infusion

SUMMARY:
Non-Hodgkin's lymphoma (NHL) is a cancer that arises from the transformation of normal B and T lymphocytes (white blood cells). The purpose of this study is to assess the safety, tolerability, pharmacokinetics, and preliminary efficacy of ABBV-291 in adult participants in relapsed or refractory (R/R) NHL, including but not limited to diffuse large b-cell lymphoma (DLBCL), mantle cell lymphoma (MCL), and follicular lymphoma (FL). Adverse events will be assessed.

ABBV-291 is an investigational drug being developed for the treatment of NHL. This study will include a dose escalation phase to determine the maximum administered dose (MAD)/Maximum tolerated dose (MTD) of ABBV-291 and a dose expansion/optimization phase to determine the change in disease activity in participants with R/R NHL. Approximately 165 adult participants with multiple NHL subtypes will be enrolled in the study in sites world wide

In the dose escalation phase of the study participants will receive escalating Intravenously (IV) infused doses of ABBV-291, until the MAD/MTD is determined. In the dose expansion/optimization phase of the study participants receive IV infused ABBV-291, as part of the approximately 74 month study duration.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, and side effects.

ELIGIBILITY:
Inclusion Criteria:

* For dose escalation (Part 1) only: Participants must have documented diagnosis of B-cell malignancies including (but not limited to) the following, with histology based on criteria established by the World Health Organization (WHO), and measurable disease requiring treatment:

  * Mantle cell lymphoma (MCL);
  * Marginal zone lymphoma (MZL);
  * Waldenstrom macroglobulinemia (WM);
  * Diffuse large b-cell lymphoma (DLBCL) (including: germinal center B-cell type, activated B-cell type, primary cutaneous DLBCL [leg type], Epstein-Barr virus-positive (EBV+) DLBCL [not otherwise specified], DLBCL associated with chronic inflammation, human herpesvirus 8-positive [HHV8+] DLBCL [not otherwise specified], B cell lymphoma [unclassifiable] with features intermediate between DLBCL and classical Hodgkin lymphoma, high-grade B-cell lymphoma [not otherwise specified], high-grade B-cell lymphoma [with MYC (avian myelocytomatosis viral oncogene homolog) and BCL2 and/or BCL6 rearrangements], DLBCL arising from follicular lymphoma [FL] [transformed FL]);
  * FL Grades 1 to 3B;
* For dose expansion (Part 2) only: Participants must have documented diagnosis of one of the following B-cell malignancies, with histology based on criteria established by the WHO, and measurable disease requiring treatment:

  * Part 2a only: DLBCL (including: germinal center B-cell type, activated B-cell type, primary cutaneous DLBCL [leg type], EBV+ DLBCL [not otherwise specified], DLBCL associated with chronic inflammation, HHV8+ DLBCL [not otherwise specified], B-cell lymphoma [unclassifiable] with features intermediate between DLBCL and classical Hodgkin lymphoma, high-grade B-cell lymphoma [not otherwise specified], high-grade B-cell lymphoma [with MYC and BCL2 and/or BCL6 rearrangements], DLBCL arising from FL [transformed FL]);
  * Part 2b only: FL Grades 1 to 3B;
  * Part 2c only: Mantle cell lymphoma;
* For all participants (Parts 1 and 2):

  * Must be considered relapsed or refractory to, or intolerant of, at least 2 or more prior lines of therapy known to provide a clinical benefit for their condition, and for whom there is no appropriate locally available therapy known to provide clinical benefit (e.g., standard chemotherapy or autologous stem cell transplantation [ASCT]).
  * Indolent non-Hodkin's lymphoma (NHL) participants must meet relevant disease specific requirements for treatment (e.g., National Comprehensive Cancer Network [NCCN], Groupe d'Etude des Lymphomes Folliculaires [GELF]).
  * History of allogeneic stem cell transplantation must be stable off of immunosuppression for at least 3 months.
  * For participants enrolled in backfill cohorts or at dose levels previously cleared, subjects must provide consent to an on-treatment fresh tumor biopsy from the same tumor lesion as the baseline tumor tissue. This requirement may be waived at the discretion of the contract research organization (CRO) Medical Monitor if collecting a biopsy would place the subject at risk of harm or would require a technically complicated procedure based on tumor location as assessed by the investigator or could hinder a subject's ability to participate in the study.
  * Previously treated with a CD79b-targeting therapy (e.g., CD79b monoclonal antibody) a core or excision tumor biopsy subsequent to the most recent CD79b-targeting therapy must be collected. Tumor biopsy requirements may be modified by Sponsor during the study. This requirement may be waived at the discretion of the contract research organization (CRO) Medical Monitor if collecting a biopsy would place the subject at risk of harm or would require a technically complicated procedure based on tumor location as assessed by the investigator or could hinder a subject's ability to participate in the study.

    * CD79b expression status will be assessed in all participants.
* Have an eastern cooperative oncology group (ECOG) Performance Status of 0 or 1.
* Laboratory values meeting the criteria in the protocol within the screening period prior to the first dose of study drug (if multiple samples are drawn within the screening period, the sample/result immediately prior to Cycle 1 Day 1 is applicable).
* Availability of representative baseline tumor tissue (most recent archived tumor tissue or fresh biopsy collected during screening phase) suitable for immunohistochemistry (IHC) testing. This requirement may be waived at the discretion of the CRO Medical Monitor if collecting a biopsy at screening would place the participant at risk of harm or would require a technically complicated procedure based on tumor location as assessed by the investigator or could hinder a participant's ability to participate in the study.

Exclusion Criteria:

* History of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids, or any evidence of active ILD or pneumonitis.
* Treatment with any of the following:

  * Anticancer therapy including chemotherapy, radiotherapy, small molecule, investigational, and biologic agents within 14 days (or at least 5 half-lives, whichever is shorter), prior to the first dose of the study treatment;
  * CD79b-directed agents (e.g., CD79b monoclonal antibody therapy) within 4 weeks (or at least 5 half-lives, whichever is shorter) prior to the first dose of study treatment.
  * Prior treatment with an antibody drug conjugate that consists of a topoisomerase I inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AE)s | Up to 74 Months
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have a causal relationship with this treatment.
Percentage of Participants with Dose Limiting Toxicities (DLT)s | Up to 74 Months
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.
Percentage of Participants with Clinically Significant Laboratory Values (Chemistry, and Hematology) | Up to 74 Months
  Percentage of participants with clinically significant laboratory values (chemistry, and hematology).
Percentage of Participants with Clinically Significant Vital Sign Measurements | Up to 74 Months
  Vital sign are defined as determinations of systolic and diastolic blood pressure, pulse rate, respiratory rate, and body temperature.
Percentage of Participants with Clinically Significant Electrocardiogram (ECG) Findings | Up to 74 Months
  Percentage of participants with clinically significant ECG findings.
Objective Response Rate (ORR) | Up to 74 Months
  ORR is defined as the percentage of participants with a confirmed best overall response (BOR) of partial response (PR) or better per disease-specific response criteria (e.g., Lugano classification).

SECONDARY OUTCOMES:
Duration of Response (DOR) as Assessed by Investigator | Up to 74 Months
  DOR is defined for participants achieving a confirmed PR or better as the time from the initial response of PR (or better) per investigator review according to disease-specific response criteria to disease progression or death of any cause, whichever occurs earlier.
Progression-Free Survival (PFS) as Assessed by Investigator | Up to 74 Months
  PFS is defined as time from first study treatment to a documented disease progression according to disease-specific response criteria, as determined by the investigator, or death due to any cause, whichever occurs earlier.
Time to response (TTR) | Up to 74 Months
  TTR is defined as time from first study treatment to the initial response of PR (or better) per investigator review according to disease-specific response criteria.
Area Under the Curve (AUC) of ABBV-291 | Up to 12 Months
  AUC is defined as the area under the plasma/serum concentration-time curve of ABBV-291.
Maximum Observed Plasma/Serum Concentration (Cmax) of ABBV-291 | Up to 12 Months
  Cmax is defined as maximum observed plasma/serum concentration of ABBV-291.
Time to Cmax (Tmax) of ABBV-291 | Up to 12 Months
  Tmax is defined as time to Cmax of ABBV-291.
Half-Life (t1/2) of ABBV-291 | Up to 12 Months
  t1/2 is defined as the half-life of ABBV-291.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (14):
- United States (5):
  - Carolina BioOncology Institute /ID# 265259, Huntersville, North Carolina
  - Willamette Valley Cancer Institute and Research Center /ID# 270945, Eugene, Oregon
  - Texas Oncology - Central/South Texas /ID# 270946, Austin, Texas
  - START Mountain Region /ID# 267592, West Valley City, Utah
  - Virginia Cancer Specialists - Fairfax /ID# 265082, Fairfax, Virginia
- Australia (2):
  - St Vincent's Hospital Melbourne /ID# 261664, Fitzroy Melbourne, Victoria
  - Sir Charles Gairdner Hospital /ID# 268579, Nedlands, Western Australia
- Israel (2):
  - Hadassah Medical Center-Hebrew University /ID# 261658, Jerusalem, Jerusalem
  - Tel Aviv Sourasky Medical Center /ID# 261659, Tel Aviv, Tel Aviv
- Japan (3):
  - Aichi Cancer Center /ID# 267471, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 261775, Kashiwa-shi, Chiba
  - The Cancer Institute Hospital Of JFCR /ID# 267470, Koto-ku, Tokyo
- United Kingdom (2):
  - The Christie /ID# 267177, Manchester
  - University Hospitals Plymouth NHS Trust /ID# 267174, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-893